CLINICAL TRIAL: NCT01800968
Title: Functional Impact of GLP-1 for Heart Failure Treatment
Brief Title: Functional Impact of GLP-1 for Heart Failure Treatment (FIGHT)
Acronym: FIGHT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00042633; 5U10HL084904-09 (NIH)
Record Dates: First submitted 2013-02-07; First posted 2013-02-28 (Estimated); Results first posted 2017-02-15 (Actual); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Acute Heart Failure
MeSH Terms: interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liraglutide (Active Comparator): Increasing dose from 0.6mg, 1.2mg to 1.8mg SQ daily.
  Interventions: Drug: Liraglutide
- Placebo (Placebo Comparator): Placebo dose increasing from 0.6mg, 1.2mg to 1.8 mg SQ daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Liraglutide — Active Drug
  Other Names: Victoza
  Arms: Liraglutide
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The primary objective is to test the hypothesis that, compared with placebo, therapy with Subcutaneous (SQ) GLP-1 agonist in the post-Acute Heart Failure Syndrome (AHFS) discharge period will be associated with greater clinical stability at six months as assessed by a composite clinical endpoint.

DETAILED DESCRIPTION:
Hospitalization for AHFS identifies individuals at increased risk of death and re-hospitalization following discharge. This increased risk justifies intervention with novel therapy during the vulnerable post-discharge period to enhance clinical stability and prevent early HF mortality and readmissions.

As heart failure (HF) progresses, impairments in metabolism render the heart substrate constrained, limiting cardiac metabolism. Glucagon-like peptide-1 (GLP-1) is a naturally occurring incretin peptide that enhances cellular glucose uptake by stimulating insulin secretion and insulin sensitivity in target tissues. Preclinical and early-phase clinical data support GLP-1 as an effective therapy for advanced HF while use of GLP-1 receptor agonists in large numbers of patients with diabetes reveal a good safety profile and reductions in adverse cardiac outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. AHFS as defined by the presence of at least 1 symptom (dyspnea, orthopnea, or edema) AND 1 sign (rales on auscultation, peripheral edema, ascites, pulmonary vascular congestion on chest radiography)
3. AHFS is the primary cause of hospitalization
4. Prior clinical diagnosis of HF
5. Left Ventricular Ejection Fraction(LVEF) ≤ 40% during the preceding 3 months (if no echo within the preceding 3 months, an LVEF ≤ 30% during the preceding three years is acceptable)
6. On evidence-based medication for HF (including beta-blocker and ACE-inhibitor/ARB) or previously deemed intolerant
7. Use of at least 80 mg or furosemide total daily dose (or equivalent) prior to admission for AHFS (a lower dose of a loop diuretic combined with a thiazide will count as an "equivalent")
8. Willingness to provide informed consent

Exclusion Criteria:

1. AHFS due to acute myocarditis or acute Myocardial Infarction
2. Ongoing hemodynamically significant arrhythmias contributing to HF decompensation
3. Inotrope, intra-aortic balloon pump (IABP) or other mechanical circulatory support use at the time of consent. Prior use will not exclude a patient.
4. Current or planned left ventricular assist device therapy in next 180 days
5. United Network for Organ Sharing status 1A or 1B
6. B-type natriuretic peptide(BNP)< 250 or NT-proBNP<1,000 (Not required per protocol but if available and too low would be an exclusion; within 48 hours of consent)
7. Hemoglobin (Hgb) < 8.0 g/dl
8. Glomerular filtration rate(GFR) < 20 ml/min/1.73 m2 within 48 hours of consent
9. Systolic blood pressure < 80 mmHg at consent
10. Resting Heart Rate > 110 at consent
11. Acute coronary syndrome within 4 weeks as defined by electrocardiographic (ECG) changes and biomarkers of myocardial necrosis (e.g. troponin) in an appropriate clinical setting (chest discomfort or anginal equivalent)
12. Percutaneous Coronary Intervention, coronary artery bypass grafting or new biventricular pacing within past 4 weeks
13. Primary hypertrophic cardiomyopathy
14. Infiltrative cardiomyopathy
15. Constrictive pericarditis or tamponade
16. Complex congenital heart disease
17. Non-cardiac pulmonary edema
18. More than moderate aortic or mitral stenosis
19. Intrinsic (prolapse, rheumatic) valve disease with severe mitral, aortic or tricuspid regurgitation
20. Sepsis, active infection (excluding cystitis) or other comorbidity driving the HF decompensation
21. Acute or chronic severe liver disease as evidenced by any of the following: encephalopathy, variceal bleeding, International Normalized Ration (INR) > 1.7 in the absence of anticoagulation treatment
22. Terminal illness (other than HF) with expected survival of less than 1 year
23. Previous adverse reaction to the study drug
24. Receipt of any investigational product in the previous 30 days.
25. Enrollment or planned enrollment in another randomized therapeutic clinical trial in next 6 months.
26. Inability to comply with planned study procedures
27. Pregnancy or breastfeeding mothers
28. Women of reproductive age not on adequate contraception
29. History of acute or chronic pancreatitis
30. History of symptomatic gastroparesis
31. Familial or personal history of medullary thyroid cancer or multiple endocrine neoplasia type-2 (MEN2)
32. Prior weight-loss surgery (i.e., Roux-en-Y gastric bypass) or other gastric surgery associated with increased endogenous GLP-1 production
33. Prior or ongoing treatment with GLP-1 receptor agonists
34. Ongoing treatment with dipeptidyl peptide-IV inhibitors (1 week washout required)
35. Ongoing treatment with thiazolidinedione
36. Oxygen-dependent chronic obstructive pulmonary disease
37. Diabetic patients with history of 2 or more severe hypoglycemia, Diabetic Ketoacidosis(DKA) or hyperglycemic, hyperosmotic nonketotic coma in the preceding 12 months.
38. Diagnosis of Type 1 Diabetes Mellitus

40. If diabetic, inadequate glycemic control with glucose level > 300 mg/dL within 24 hours of randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2013-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Hernandez, MD, Principal Investigator — Duke University; Eugene Bruanwald, MD, Study Chair — Harvard University
Locations (25):
- United States (25):
  - Christiana Care Health Services, Newark, Delaware
  - Emory University School of Medicine, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston VA Healtcare System, West Roxbury, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Saint Louis University Hospital, St Louis, Missouri
  - Duke University, Durham, North Carolina
  - Southeast Regional Medical Center, Lumberton, North Carolina
  - University Hospitals- Case Medical Center, Cleveland, Ohio
  - Metro Health System, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Lancaster Heart and Stroke Foundation, Lancaster, Pennsylvania
  - University of Pennsylvaina, Philadelphia, Pennsylvania
  - Jefferson Medical College, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Michael Debakey VA Medical Center, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Utah School of Medicine, Salt Lake City, Utah
  - Utah VA Medical Center, Salt Lake City, Utah
  - The University of Vermont- Fletcher Allen Health Care, Burlington, Vermont

REFERENCES:
- [Derived] Lerman JB, Giamberardino SN, Hernandez AF, Felker GM, Shah SH, McGarrah RW. Plasma metabolites associated with functional and clinical outcomes in heart failure with reduced ejection fraction with and without type 2 diabetes. Sci Rep. 2022 Jun 2;12(1):9183. doi: 10.1038/s41598-022-12973-0. PMID 35654972
- [Derived] Redouane B, Greene SJ, Fudim M, Vaduganathan M, Ambrosy AP, Sun JL, DeVore AD, McNulty SE, Mentz RJ, Hernandez AF, Felker GM, Cooper LB, Borlaug BA, Velazquez EJ, Margulies KB, Sharma A. Effects of Liraglutide on Worsening Renal Function Among Patients With Heart Failure With Reduced Ejection Fraction: Insights From the FIGHT Trial. Circ Heart Fail. 2020 May;13(5):e006758. doi: 10.1161/CIRCHEARTFAILURE.119.006758. Epub 2020 May 4. PMID 32362166
- [Derived] Sharma A, Ambrosy AP, DeVore AD, Margulies KB, McNulty SE, Mentz RJ, Hernandez AF, Michael Felker G, Cooper LB, Lala A, Vader J, Groake JD, Borlaug BA, Velazquez EJ. Liraglutide and weight loss among patients with advanced heart failure and a reduced ejection fraction: insights from the FIGHT trial. ESC Heart Fail. 2018 Dec;5(6):1035-1043. doi: 10.1002/ehf2.12334. Epub 2018 Aug 17. PMID 30120812
- [Derived] Margulies KB, Hernandez AF, Redfield MM, Givertz MM, Oliveira GH, Cole R, Mann DL, Whellan DJ, Kiernan MS, Felker GM, McNulty SE, Anstrom KJ, Shah MR, Braunwald E, Cappola TP; NHLBI Heart Failure Clinical Research Network. Effects of Liraglutide on Clinical Stability Among Patients With Advanced Heart Failure and Reduced Ejection Fraction: A Randomized Clinical Trial. JAMA. 2016 Aug 2;316(5):500-8. doi: 10.1001/jama.2016.10260. PMID 27483064

RESULTS

PARTICIPANT FLOW:
Groups:
- Liraglutide: Increasing dose from 0.6mg, 1.2mg to 1.8mg subcutaneous daily.
  Liraglutide: Active Drug
- Placebo: Placebo dose increasing from 0.6mg, 1.2mg to 1.8 mg subcutaneous daily.
  Placebo: Placebo
Period: Overall Study
Arm/Group | Liraglutide | Placebo
Started | 154 | 146
Completed | 118 | 114
Not Completed | 36 | 32
Not completed — Death | 23 | 16
Not completed — Lost to Follow-up | 5 | 7
Not completed — Withdrawal by Subject | 7 | 9
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: All patients randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Liraglutide | Placebo | Total
Number analyzed (Participants) | 154 | 146 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (12.9) | 59.6 (12.2) | 59.7 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 33 | 64
  Male | 123 | 113 | 236
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 11 | 15
  Not Hispanic or Latino | 150 | 135 | 285
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 3 | 7
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 67 | 48 | 115
  White | 82 | 90 | 172
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Global Ranking of Predefined Events
Description: A rank score based on time to death, time to adjudicated heart failure hospitalization, and time-averaged proportional change in NTproBNP through d180. For patients that died, the patient with the shortest time from randomization to death is assigned rank 1, the second shortest time is assigned rank 2, etc. The patient with the longest time from randomization to death is assigned rank X. For patients that did not die but had a heart failure hospitalization, the patient with the shortest time from randomization to re-admission is assigned rank X+1 and the patient with the longest time from randomization to heart failure hospitalization is assigned rank Y. For patients that did not die or have a heart failure hospitalization, increases in time-averaged proportional change in NTproBNP indicate a worse result and the largest increase is assigned rank Y+1. The patient with the largest decrease is assigned rank N, where N is the sample size.
Time Frame: Randomization to 180 days
Population: All randomized subjects.
Measure: Mean (Standard Deviation); unit: rank
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 154 | 146
rank | 145.5 (88.1) | 155.7 (85.3)
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; Test type: Superiority or Other; p = 0.3087, Rank score

2. Secondary Outcome: Change in Left Ventricular End-Diastolic Volume Index
Description: Change in Left Ventricular End-Diastolic Volume Index from baseline to 180 days.
Time Frame: Baseline to 180 days
Population: All randomized subjects.
Measure: Mean (Standard Deviation); unit: ml per meter squared
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 154 | 146
ml per meter squared | 3.37 (31.9) | -2.91 (32.04)
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; Test type: Superiority or Other; p = 0.1549, Regression, Linear

3. Secondary Outcome: Change in Left Ventricular End-systolic Volume Index
Description: Change in left ventricular end-systolic volume index from baseline to day 180.
Time Frame: Baseline to 180 days
Population: All randomized subjects.
Measure: Mean (Standard Deviation); unit: ml per meter squared
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 154 | 146
ml per meter squared | 1.16 (26.2) | -3.47 (26.5)
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; Test type: Superiority or Other; p = 0.1932, Regression, Linear

4. Secondary Outcome: Change in Left Ventricular Ejection Fraction
Description: Change in left ventricular ejection fraction from baseline to day 180
Time Frame: Baseline to 180 days
Population: All randomized subjects.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 154 | 146
percent | 1.07 (9.1) | 1.37 (10.0)
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; Test type: Superiority or Other; p = 0.9535, Regression, Linear

5. Secondary Outcome: Change in Medial Filling Pressure
Description: Change in medial filling pressure baseline to day 180.
Time Frame: Baseline to 180 days
Population: All randomized subjects.
Measure: Mean (Standard Deviation); unit: m/sec
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 154 | 146
m/sec | 1.12 (18.8) | 0.25 (17.8)
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; Test type: Superiority or Other; p = 0.8548, Regression, Linear

6. Secondary Outcome: Change in Lateral Filling Pressure
Description: Change in lateral filling pressure baseline to day 180.
Time Frame: Baseline to 180 days
Population: All randomized subjects.
Measure: Mean (Standard Deviation); unit: m/sec
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 154 | 146
m/sec | -0.05 (12.3) | 0.39 (13.1)
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; Test type: Superiority or Other; p = 0.4266, Regression, Linear

7. Secondary Outcome: Change in 6 Minute Walk Distance
Description: Change in 6 minute walk distance baseline to day 30
Time Frame: Baseline to day 30
Population: All randomized subjects.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 154 | 146
meters | 50.4 (110.8) | 37.3 (99.6)
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; Test type: Superiority or Other; p = 0.1705, Regression, Linear

8. Secondary Outcome: Change in 6 Minute Walk Distance
Description: Change in 6 minute walk distance baseline to 90 days.
Time Frame: Baseline to 90 days
Population: All randomized subjects.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 154 | 146
meters | 56.8 (132.7) | 38.7 (115.4)
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; Test type: Superiority or Other; p = 0.1309, Regression, Linear

9. Secondary Outcome: Change in 6 Minute Walk Distance
Description: Change in 6 minute walk distance baseline to 180 days.
Time Frame: Baseline to 180 days
Population: All randomized subjects.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 154 | 146
meters | 55.7 (133.9) | 55.3 (127.2)
Statistical Analysis 1: Comparison: Liraglutide; Test type: Superiority or Other; p = 0.7920, Regression, Linear

10. Secondary Outcome: Change in Clinical Summary Score Using the Kansas City Cardiomyopathy Questionnaire (KCCQ)
Description: Change in clinical summary score using the Kansas City Cardiomyopathy Questionnaire (KCCQ) baseline to 30 days. The Kansas City Cardiomyopathy Questionnaire is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life.In the KCCQ, an overall summary score can be derived from the physical function, symptom (frequency and severity), social function and quality of life domains. For each domain, the validity, reproducibility, responsiveness and interpretability have been independently established. Each question is answered by the subject on a 6 point scale (Extremely limited, quite a bit limited, moderately limited, slightly limited, not at all limited, Limited for other reasons or did not do this activity).Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Time Frame: Baseline to 30 days
Population: All randomized subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 154 | 146
units on a scale | 14.69 (25.90) | 14.44 (22.03)
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; Test type: Superiority or Other; p = 0.7026, Regression, Linear

11. Secondary Outcome: Change in Clinical Summary Score Using the Kansas City Cardiomyopathy Questionnaire (KCCQ)
Description: Change in clinical summary score using the Kansas City Cardiomyopathy Questionnaire (KCCQ) baseline to 90 days.The Kansas City Cardiomyopathy Questionnaire is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life.In the KCCQ, an overall summary score can be derived from the physical function, symptom (frequency and severity), social function and quality of life domains. For each domain, the validity, reproducibility, responsiveness and interpretability have been independently established. Each question is answered by the subject on a 6 point scale (Extremely limited, quite a bit limited, moderately limited, slightly limited, not at all limited, Limited for other reasons or did not do this activity).Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Time Frame: Baseline to 90 days
Population: All randomized subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 154 | 146
units on a scale | 13.86 (24.99) | 11.72 (23.82)
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; Test type: Superiority or Other; p = 0.2662, Regression, Linear

12. Secondary Outcome: Change in Clinical Summary Score Using the Kansas City Cardiomyopathy Questionnaire (KCCQ)
Description: Change in clinical summary score using the Kansas City Cardiomyopathy Questionnaire (KCCQ) from baseline to day 180.The Kansas City Cardiomyopathy Questionnaire is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life.In the KCCQ, an overall summary score can be derived from the physical function, symptom (frequency and severity), social function and quality of life domains. For each domain, the validity, reproducibility, responsiveness and interpretability have been independently established. Each question is answered by the subject on a 6 point scale (Extremely limited, quite a bit limited, moderately limited, slightly limited, not at all limited, Limited for other reasons or did not do this activity).Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Time Frame: Baseline to day 180
Population: All randomized subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 154 | 146
units on a scale | 13.79 (23.83) | 13.14 (23.60)
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; Test type: Superiority or Other; p = 0.6395, Regression, Linear

13. Secondary Outcome: Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) Overall Summary Score
Description: Kansas City Cardiomyopathy Questionnaire (KCCQ) change in overall summary score baseline to 30 days.The Kansas City Cardiomyopathy Questionnaire is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life.In the KCCQ, an overall summary score can be derived from the physical function, symptom (frequency and severity), social function and quality of life domains. For each domain, the validity, reproducibility, responsiveness and interpretability have been independently established. Each question is answered by the subject on a 6 point scale (Extremely limited, quite a bit limited, moderately limited, slightly limited, not at all limited, Limited for other reasons or did not do this activity).Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Time Frame: Baseline to 30 days
Population: All randomized subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 154 | 146
units on a scale | 12.98 (23.82) | 14.01 (20.09)
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; Test type: Superiority or Other; p = 0.8218, Regression, Linear

14. Secondary Outcome: Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) Overall Summary Score
Description: Kansas City Cardiomyopathy Questionnaire (KCCQ) change in overall summary score baseline to 90 days.The Kansas City Cardiomyopathy Questionnaire is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life.In the KCCQ, an overall summary score can be derived from the physical function, symptom (frequency and severity), social function and quality of life domains. For each domain, the validity, reproducibility, responsiveness and interpretability have been independently established. Each question is answered by the subject on a 6 point scale (Extremely limited, quite a bit limited, moderately limited, slightly limited, not at all limited, Limited for other reasons or did not do this activity).Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Time Frame: Baseline to 90 days
Population: All randomized subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 154 | 146
units on a scale | 14.17 (24.46) | 10.62 (22.48)
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; Test type: Superiority or Other; p = 0.1124, Regression, Linear

15. Secondary Outcome: Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) Overall Summary Score.
Description: Kansas City Cardiomyopathy Questionnaire (KCCQ) change in overall summary score baseline to 180 days.The Kansas City Cardiomyopathy Questionnaire is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life.In the KCCQ, an overall summary score can be derived from the physical function, symptom (frequency and severity), social function and quality of life domains. For each domain, the validity, reproducibility, responsiveness and interpretability have been independently established. Each question is answered by the subject on a 6 point scale (Extremely limited, quite a bit limited, moderately limited, slightly limited, not at all limited, Limited for other reasons or did not do this activity).Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Time Frame: Baseline to 180 days
Population: All randomized subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 154 | 146
units on a scale | 13.44 (22.61) | 13.25 (22.38)
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; Test type: Superiority or Other; p = 0.8088, Regression, Linear

16. Secondary Outcome: Individual Component of the Primary Endpoint- Mortality
Description: Individual component of the primary endpoint of mortality at 180 days after randomization
Time Frame: Randomization to 180 days
Population: All randomized subjects.
Measure: Number; unit: participants
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 154 | 146
participants | 19 | 16
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; Test type: Superiority or Other; p = 0.7764, Log Rank

17. Secondary Outcome: Individual Component of the Primary Endpoint- Heart Failure Hospitalization
Description: Individual component of the primary endpoint- Heart Failure hospitalization from randomization to 180 days
Time Frame: Randomization to 180 days
Population: All randomized subjects.
Measure: Number; unit: participants
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 154 | 146
participants | 63 | 50
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; Test type: Superiority or Other; p = 0.1701, Log Rank

18. Secondary Outcome: Individual Component of the Primary Endpoint- Time-averaged Proportional Change in NT-proBNP
Description: Individual component of the primary endpoint- time-averaged proportional change in NT-proBNP from baseline to 180 days
Time Frame: Baseline to 180 days
Population: All randomized subjects.
Measure: Mean (Standard Deviation); unit: weighted average of ratio to baseline
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 154 | 146
weighted average of ratio to baseline | 335.81 (445.8) | 317 (307.64)
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; Test type: Superiority or Other; p = 0.6532, Regression, Linear

19. Secondary Outcome: Global Ranking of Predefined Events
Description: A rank score based on time to death, time to adjudicated heart failure hospitalization, time to emergency department visit and time-averaged proportional change in NTproBNP through d180. See Outcome Measure 1 for a general description of the outcome derivation.
Time Frame: Baseline to 180 days
Population: All randomized subjects.
Measure: Mean (Standard Deviation); unit: rank
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 154 | 146
rank | 144.29 (87.63) | 157.05 (85.61)
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; Test type: Superiority or Other; p = 0.2033, Rank score

ADVERSE EVENTS:
Time Frame: Baseline to day 210.
Description: All serious adverse events documented from baseline to day 210. According to protocol: Non-serious adverse events will not be collected on the eCRF but should be documented in source documents and followed according to local standard of care. Non-serious adverse events were not reported to sponsor, and therefore not reported.
Groups:
- Liraglutide: Increasing dose from 0.6mg, 1.2mg to 1.8mg subcutaneous (SQ) daily.
  Liraglutide: Active Drug
- Placebo: Placebo dose increasing from 0.6mg, 1.2mg to 1.8 mg subcutaneous (SQ) daily.
  Placebo: Placebo
Arm/Group | Liraglutide | Placebo
Serious Adverse Events (participants affected / at risk) | 33/154 | 33/146
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide (N=154) | Placebo (N=146)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Angina pectoris (Cardiac disorders) | 2 (3) | 0 (0)
Gastrointentinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 3 (3)
Non-cardiac chest pain (General disorders) | 2 (2) | 1 (1)
Diverticulitis (Infections and infestations) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 4 (4) | 3 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hepatic Encephalopathy (Nervous system disorders) | 2 (2) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 4 (4) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 4 (5)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
International Normalised Ratio Increased (Investigations) | 2 (2) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hernia (General disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Viral Rash (Infections and infestations) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hyperolmolar Hyperglycaemic State (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hypoglycaemic unconsciousness (Nervous system disorders) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No